CLINICAL TRIAL: NCT00679601
Title: An Open-label, Multiple-dose Study Of The Absorption And Systemic Pharmacokinetics Of An2690 Applied As A 7.5% Solution To All Toenails Of Adult Patients With Moderate To Severe Onychomycosis
Brief Title: Absorption and Systemic Study of AN2690 in Patients With Moderate to Severe Onychomycosis (ADME II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: AN2690-ONYC-205; C3371014 (Other: Alias Study Number)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Fungal Nail
MeSH Terms: conditions — Onychomycosis | interventions — tavaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AN2690 — AN2690 7.5% Solution, once daily for 28 days

SUMMARY:
The purpose of the study is to determine the absorption and systemic pharmacokinetics of AN2690 following daily application to all ten (10) toenails for 28 days.

DETAILED DESCRIPTION:
A single center, open-label, multiple-dose study design will be used. Planned enrollment is 20 subjects to complete 15. Subjects must have a clinical diagnosis of onychomycosis of each great toenail and a clinical diagnosis of onychomycosis of six of the remaining toenails.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤65
* BMI between 18.5 and 35 inclusive
* Moderate to severe onychomycosis involving ≥80% of both great toenails, as determined by visual inspection after the nail has been trimmed
* Combined thickness of the nail plate and nail bed of each great toenail is >3mm
* At least 6 additional toenails with a clinical diagnosis of onychomycosis
* If a female of childbearing potential, must be using of a highly effective method of birth control or abstinence and be willing to remain on that same method of birth control throughout the study
* Capable of understanding and signing the informed consent, and willing to comply with all requirements of the study

Exclusion Criteria:

* History of allergy to any of the study drug or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure
* Clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his/her safety
* Diabetes mellitus requiring treatment other than diet and exercise
* Willing to refrain from the use of nail cosmetics such as clear and or colored nail lacquers from the screening visit until the end of the study
* Nursing, pregnant or planning to become pregnant during the study
* Failure to complete the specified washout period(s) for the following topical:

  1. Topical antifungal applied to the feet (does not include antifungals for treatment of T. pedis during the study): 4 weeks
  2. Anti-inflammatories, corticosteroids, topical immunomodulators: 2 weeks
* Failure to complete the specified washout period(s) for the following systemic medications:

  1. Corticosteroids (including intramuscular injections): 2 weeks
  2. Antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophyte: 24 weeks
  3. Systemic immunomodulators: 4 weeks
* Received treatment of any type for cancer within the last 6 months
* History of any significant internal disease
* Nail or anatomic abnormalities of the toe, e.g., genetic nail disorders, primentary disorders, onychogryphosis, trauma to the nail(s) to be treated
* AIDS or AIDS related complex
* History of street drug or alcohol abuse
* Donated or lost blood, or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six-week period preceding study initiation
* Donated plasma during the two week period preceding study initiation
* Participated in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study
* Prior enrollment in a study using the study drug, AN2690

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03-31 (Actual); Primary Completion 2007-05-31 (Actual); Study Completion 2007-05-31 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of AN2690 in plasma and the concentration of AN2690 in urine over time | Days 0, 1, 14, 15, and 28

SECONDARY OUTCOMES:
Efficacy measures of linear toenail growth, fungal culture results, KOH results, and clear toenail growth | Days 0, 14, 28, and 42
Safety and tolerance assessed by application site reactions, adverse events, vital signs, physical examinations, and 12-lead EKG | Days 0-28, and 42

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- J&S Studies, Bryan, Texas, United States